CLINICAL TRIAL: NCT05602337
Title: A Prospective Multicenter Sample Collection Study Using Non-invasive Methods to Investigate Mutation Burden in Non-lesional Facial Skin of Patients With a History of Skin Cancer
Brief Title: A Prospective Multicenter Sample Collection Study Using Non-invasive Methods to Investigate Mutation Burden in Non-lesional Facial Skin of Patients With a Hx of Skin Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: DermTech (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: DermTech 2022
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Melanoma and Other Malignant Neoplasms of Skin
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Non-invasively collected skins samples will be harvested with adhesive patches and stored for batch analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Immunocompetent BCC Subjects: BCC-predominant group
  Interventions: Other: Observational Study Only
- Immunocompetent SCC Subjects: SCC-predominant group
  Interventions: Other: Observational Study Only
- Immunocompetent MM Subjects: Melanoma group
  Interventions: Other: Observational Study Only
- Control: age, sex and Fitzpatrick phototype match
  Interventions: Other: Observational Study Only
- Solid Organ Transplantation Recipient - SC: At least 5 skin cancers and at least 5 years post-transplant
  Interventions: Other: Observational Study Only
- Solid Organ Transplantation Recipient: No more than 1 skin cancer and at least 5 years post-transplant
  Interventions: Other: Observational Study Only

INTERVENTIONS:
Other: Observational Study Only — Non-invasive Skin Sampling
  Other Names: Non-invasive Skin Sampling

SUMMARY:
This is a prospective, multicenter, sample collection study using DermTech's non-invasive skin collection kits to evaluate the mutation burden of non-lesional facial skin from subjects with a documented history of numerous basal cell carcinomas, squamous cell carcinomas or melanomas compared to that of subjects with no history of skin cancer matched for age, sex and Fitzpatrick phototype.

DETAILED DESCRIPTION:
This is a prospective, multicenter, sample collection study using DermTech's non-invasive skin collection kits to evaluate the mutation burden of non-lesional facial skin from subjects with a documented history of numerous basal cell carcinomas, squamous cell carcinomas or melanomas compared to that of subjects with no history of skin cancer matched for age, sex and Fitzpatrick phototype.

Approximately 20-30 participants will be enrolled in each of six (6) main groups outlined below for a total of 120-180 subjects and controls:

ELIGIBILITY:
Inclusion Criteria:

For the immunocompetent (non-SOTR) groups, a subject will be eligible if he or she:

1. Is at least 18 years of age;
2. Is willing to consent to non-invasive adhesive tape sampling and DNA mutation burden analysis;
3. Has a history of 10 or more basal cell carcinomas (BCCs) and at least a 10:1 ratio of BCC to other skin cancer types; or
4. Has a history of 5 or more squamous cell carcinomas (SCCs) and at least a 5:1 ratio of SCC to other skin cancer types; or
5. Has a history of 3 or more melanomas; or

   For the immunocompetent controls:
6. Has no history of skin cancer but is an age, birth sex, and Fitzpatrick phototype match (control) for an enrolled participant.

   For the SOTR groups, a subject will be eligible if he or she:
7. Is age 50-70;
8. Received a heart, lung, kidney, or liver transplant at least 5 years prior to study enrollment; or
9. Has a history of 5 or more keratinocyte carcinomas (BCC or SCC), or a history of 3 or more melanomas following organ transplantation.

   For the SOTR controls:
10. Is a transplant recipient age 50-70 with no more than 2 keratinocyte carcinomas.

Exclusion Criteria:

1. Has applied certain topical medications (corticosteroids, alpha-hydroxy acids, retinoids, antibiotics, etc.) to the skin to be sampled within 30 days of beginning the study;
2. Has undergone field therapy for actinic keratoses (e.g. 5-fluorouracil) involving the skin to be sampled within the past 12 months;
3. Has a generalized skin disorder not related to skin cancer such as psoriasis, photosensitivity disorder, or eczematous dermatitis affecting the skin to be sampled;
4. Has a known allergy to latex rubber or tape adhesives;
5. Is currently participating in another investigational study, or has participated in another study within 30 days of initiating the current study;
6. Has applied a sunscreen, moisturizer, or other topical to the skin to be sampled that cannot be adequately removed and may therefore compromise sample collection;
7. Has clinical findings which the Investigator determines may put the subject at undue risk or may interfere with the study;
8. Has undergone phototherapy or used a tanning bed within 3 months of beginning the study;
9. Has used systemic retinoids, chemotherapeutics, or immunotherapy within 3 months of beginning the study;
10. Has used an immunosuppressive medication within 3 months of study initiation, such as azathioprine, cyclosporine, methotrexate, or any of the immunosuppressive biological therapies (TNF-inhibitors, etc.);
11. Is known or suspected to have a cancer predisposition syndrome (CPS), such as Gorlin syndrome / basal cell nevus syndrome, Xeroderma pigmentosum, Ferguson-Smith syndrome, Oculocutaneous albinism, Epidermolysis bullosa, Epidermodysplasia verruciformis, Fanconi anemia, Rombo syndrome, Bazex-Dupre-Christol syndrome, Bloom syndrome, Werner syndrome, Dyskeratosis congenita, Hereditary Breast and Ovarian Cancer (HBOC) syndrome, Lynch syndrome, etc.;
12. Is known or suspected to harbor a pathogenic germline mutation within one or more cancer predisposition genes, such as TP53, CDKN2A, NF1, BAP1, DICER1, FH, SDHD, VHL, etc.; and
13. Has a history of skin cancer that cannot be verified.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Immunocompetent subjects:
  1. BCC-predominant group: Subjects with a history of 10 or more basal cell carcinomas (BCCs) and at least a 10:1 ratio of BCC to other skin cancer types
  2. SCC-predominant group: Subjects with a history of 5 or more squamous cell carcinomas (SCC) and at least a 5:1 ratio of SCC to other skin cancer types
  3. Melanoma group: Subjects with at least 3 melanomas (invasive or in situ)
  4. Control group: Sex, age (50-70 years) and Fitzpatrick phototype-matched controls
     SOTR subjects:
  5. Solid-organ transplant recipients (SOTR) with a history of at least 5 skin cancers, who are age 50-70 and at least 5-years post-transplant
  6. Solid-organ transplant recipients with no more than 1 skin cancer, who are age 50-70 years and at least 5-years post-transplant
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate genomic changes associated with increased risk of skin cancers | 1- year
  Non-invasively assess skin samples collected from facial skin from participants with a history of non-melanoma skin cancers and melanoma skin cancer compared to age, sex and Fitzpatrick phototype controls

SECONDARY OUTCOMES:
Evaluate the potential differences in the number and/or type of mutations in non-lesional skin in solid organ transplant recipients | 1-year
  Non-invasively assess skin samples collected from facial skin from solid organ transplant recipients.

CONTACTS AND LOCATIONS:
Overall Officials: James Rock, Study Director — DermTech
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided